CLINICAL TRIAL: NCT02865434
Title: An Evaluation of the Safety of Escalating Doses of Tc 99m Tilmanocept by Intravenous (IV) Injection and Skeletal Joint Imaging With SPECT in Subjects With Active Rheumatoid Arthritis (RA) and Healthy Controls
Brief Title: Evaluating Safety of Escalating Doses of Tilmanocept by IV Injection and SPECT Imaging in Subjects With and Without RA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-21
Record Dates: First submitted 2016-08-05; First posted 2016-08-12 (Estimated); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- Group 1 (RA) (Experimental): Group 1 will receive 50 µg Tc99m-tilmanocept radiolabeled with 10 mCi Tc99m as a single IV injection. Subjects will receive SPECT Imaging (60 Minutes post-injection) and SPECT Imaging (180 Minutes post-injection).
  Interventions: Drug: Tc99m-tilmanocept; Procedure: SPECT Imaging (60 Minutes post-injection); Procedure: SPECT Imaging (180 Minutes post-injection); Procedure: Planar Image with both Hands in Field of View
- Group 2 (RA) (Experimental): Group 2 will receive 200 µg Tc99m-tilmanocept radiolabeled with 10 mCi Tc99m via IV injection. Subjects will receive SPECT Imaging (60 Minutes post-injection) and SPECT Imaging (180 Minutes post-injection).
  Interventions: Drug: Tc99m-tilmanocept; Procedure: SPECT Imaging (60 Minutes post-injection); Procedure: SPECT Imaging (180 Minutes post-injection); Procedure: Planar Image with both Hands in Field of View
- Group 3 (RA) (Experimental): Group 3 will receive 400 µg Tc99m-tilmanocept radiolabeled with 10 mCi Tc99m via IV injection. Subjects will receive SPECT Imaging (60 Minutes post-injection) and SPECT Imaging (180 Minutes post-injection).
  Interventions: Drug: Tc99m-tilmanocept; Procedure: SPECT Imaging (60 Minutes post-injection); Procedure: SPECT Imaging (180 Minutes post-injection); Procedure: Planar Image with both Hands in Field of View
- Group 4 (RA) (Experimental): Group 4 will receive 50 µg Tc99m-tilmanocept radiolabeled with 5 mCi Tc99m via IV injection. Subjects will receive SPECT Imaging (60 Minutes post-injection) and SPECT Imaging (180 Minutes post-injection).
  Interventions: Drug: Tc99m-tilmanocept; Procedure: SPECT Imaging (60 Minutes post-injection); Procedure: SPECT Imaging (180 Minutes post-injection); Procedure: Planar Image with both Hands in Field of View
- Group 5 (RA) (Experimental): Group 5 will receive 200 µg Tc99m-tilmanocept radiolabeled with 5 mCi Tc99m via IV injection. Subjects will receive SPECT Imaging (60 Minutes post-injection) and SPECT Imaging (180 Minutes post-injection).
  Interventions: Drug: Tc99m-tilmanocept; Procedure: SPECT Imaging (60 Minutes post-injection); Procedure: SPECT Imaging (180 Minutes post-injection); Procedure: Planar Image with both Hands in Field of View
- Group 6 (RA) (Experimental): Group 6 will receive 400 µg Tc99m-tilmanocept radiolabeled with 5 mCi Tc99m via IV injection. Subjects will receive SPECT Imaging (60 Minutes post-injection) and SPECT Imaging (180 Minutes post-injection).
  Interventions: Drug: Tc99m-tilmanocept; Procedure: SPECT Imaging (60 Minutes post-injection); Procedure: SPECT Imaging (180 Minutes post-injection); Procedure: Planar Image with both Hands in Field of View
- Group 7 (RA) (Experimental): Group 7 will receive 50 µg Tc99m-tilmanocept radiolabeled with 1 mCi Tc99m via IV injection. Subjects will receive SPECT Imaging (60 Minutes post-injection) and SPECT Imaging (180 Minutes post-injection).
  Interventions: Drug: Tc99m-tilmanocept; Procedure: SPECT Imaging (60 Minutes post-injection); Procedure: SPECT Imaging (180 Minutes post-injection); Procedure: Planar Image with both Hands in Field of View
- Group 8 (RA) (Experimental): Group 8 will receive 200 µg Tc99m-tilmanocept radiolabeled with 1 mCi Tc99m via IV injection. Subjects will receive SPECT Imaging (60 Minutes post-injection) and SPECT Imaging (180 Minutes post-injection).
  Interventions: Drug: Tc99m-tilmanocept; Procedure: SPECT Imaging (60 Minutes post-injection); Procedure: SPECT Imaging (180 Minutes post-injection); Procedure: Planar Image with both Hands in Field of View
- Group 9 (RA) (Experimental): Group 9 will receive 400 µg Tc99m-tilmanocept radiolabeled with 1 mCi Tc99m via IV injection. Subjects will receive SPECT Imaging (60 Minutes post-injection) and SPECT Imaging (180 Minutes post-injection).
  Interventions: Drug: Tc99m-tilmanocept; Procedure: SPECT Imaging (60 Minutes post-injection); Procedure: SPECT Imaging (180 Minutes post-injection); Procedure: Planar Image with both Hands in Field of View
- Group 10 (Healthy Controls) (Experimental): Group 10 will receive Tc99m-tilmanocept at the MTD via IV injection, Whole body planar SPECT imaging (15 Minutes post-injection) , Whole body planar SPECT imaging (60 minutes post-injection) , Whole body planar SPECT imaging (180 minutes post-injection), and Whole body planar SPECT imaging (18-20 hours post-injection), Planar Image with both Hands in Field of View (60 minutes and 180 minutes post-injection), Blood Collection for PK Testing (15 Mins Before Injection), Blood Collection for PK Testing (after Injection) , Blood Collection for PK Testing (15 minutes post injection) , Blood Collection for PK Testing (60 minutes post injection) , Blood Collection for PK Testing (180 minutes post injection) , and Blood Collection for PK Testing (18-20 hours post injection).
  Interventions: Procedure: Whole body planar SPECT imaging (15 Minutes post-injection); Procedure: Whole body planar SPECT imaging (60 Minutes post-injection); Procedure: Whole body planar SPECT imaging (180 Minutes post-injection); Procedure: Whole body planar SPECT imaging (18-20 Hours post-injection); Procedure: Blood Collection for PK Testing (15 Mins Before Injection); Procedure: Blood Collection for PK Testing (after injection); Procedure: Blood Collection for PK Testing (15 minutes post injection); Procedure: Blood Collection for PK Testing (60 minutes post injection); Procedure: Blood Collection for PK Testing (180 minutes post injection); Procedure: Blood Collection for PK Testing (18-20 hours post injection); Procedure: Planar Image with both Hands in Field of View
- Group 11 (RA) (Experimental): Group 11 will receive Tc99m-tilmanocept at the MTD via IV injection, Whole body planar SPECT imaging (15 Minutes post-injection) , Whole body planar SPECT imaging (60 minutes post-injection) , Whole body planar SPECT imaging (180 minutes post-injection), and Whole body planar SPECT imaging (18-20 hours post-injection), Planar Image with both Hands in Field of View (60 minutes and 180 minutes post-injection), Blood Collection for PK Testing (15 Mins Before Injection), Blood Collection for PK Testing (after Injection) , Blood Collection for PK Testing (15 minutes post injection) , Blood Collection for PK Testing (60 minutes post injection) , Blood Collection for PK Testing (180 minutes post injection) , and Blood Collection for PK Testing (18-20 hours post injection).
  Interventions: Procedure: Whole body planar SPECT imaging (15 Minutes post-injection); Procedure: Whole body planar SPECT imaging (60 Minutes post-injection); Procedure: Whole body planar SPECT imaging (180 Minutes post-injection); Procedure: Whole body planar SPECT imaging (18-20 Hours post-injection); Procedure: Blood Collection for PK Testing (15 Mins Before Injection); Procedure: Blood Collection for PK Testing (after injection); Procedure: Blood Collection for PK Testing (15 minutes post injection); Procedure: Blood Collection for PK Testing (60 minutes post injection); Procedure: Blood Collection for PK Testing (180 minutes post injection); Procedure: Blood Collection for PK Testing (18-20 hours post injection); Procedure: Planar Image with both Hands in Field of View

INTERVENTIONS:
Drug: Tc99m-tilmanocept — Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Other Names: tilmanocept
  Arms: Group 1 (RA); Group 2 (RA); Group 3 (RA); Group 4 (RA); Group 5 (RA); Group 6 (RA); Group 7 (RA); Group 8 (RA); Group 9 (RA)
Procedure: SPECT Imaging (60 Minutes post-injection) — Subjects enrolled in Groups 1-9 will receive whole body planar SPECT imaging with 3D SPECT or SPECT/CT for targeted joints of interest 60 Minutes post-injection.
  Arms: Group 1 (RA); Group 2 (RA); Group 3 (RA); Group 4 (RA); Group 5 (RA); Group 6 (RA); Group 7 (RA); Group 8 (RA); Group 9 (RA)
Procedure: SPECT Imaging (180 Minutes post-injection) — Subjects enrolled in Groups 1-9 will receive whole body planar SPECT imaging with 3D SPECT or SPECT/CT for targeted joints of interest 180 Minutes post-injection.
  Arms: Group 1 (RA); Group 2 (RA); Group 3 (RA); Group 4 (RA); Group 5 (RA); Group 6 (RA); Group 7 (RA); Group 8 (RA); Group 9 (RA)
Procedure: Whole body planar SPECT imaging (15 Minutes post-injection) — Subjects enrolled in Groups 10-11 will receive a whole body planar SPECT scan performed 15 minutes post-injection for dosimetry.
  Arms: Group 10 (Healthy Controls); Group 11 (RA)
Procedure: Whole body planar SPECT imaging (60 Minutes post-injection) — Subjects enrolled in Groups 10-11 will receive a whole body planar SPECT scan performed 60 minutes post-injection for dosimetry.
  Arms: Group 10 (Healthy Controls); Group 11 (RA)
Procedure: Whole body planar SPECT imaging (180 Minutes post-injection) — Subjects enrolled in Groups 10-11 will receive a whole body planar SPECT scan performed 180 minutes post-injection for dosimetry.
  Arms: Group 10 (Healthy Controls); Group 11 (RA)
Procedure: Whole body planar SPECT imaging (18-20 Hours post-injection) — Subjects enrolled in Groups 10-11 will receive a whole body planar SPECT scan performed 18-20 Hours post-injection for dosimetry.
  Arms: Group 10 (Healthy Controls); Group 11 (RA)
Procedure: Blood Collection for PK Testing (15 Mins Before Injection) — Blood will be collected for subjects enrolled in Groups 10-11 for the purpose of PK analysis within 15 minutes prior to administration of Tc 99m tilmanocept
  Arms: Group 10 (Healthy Controls); Group 11 (RA)
Procedure: Blood Collection for PK Testing (after injection) — Blood will be collected for subjects enrolled in Groups 10-11 for the purpose of PK analysis immediately following administration of Tc 99m tilmanocept (00:00)
  Arms: Group 10 (Healthy Controls); Group 11 (RA)
Procedure: Blood Collection for PK Testing (15 minutes post injection) — Blood will be collected for subjects enrolled in Groups 10-11 for the purpose of PK analysis at 15 ± 5 minutes post injection of Tc 99m tilmanocept
  Arms: Group 10 (Healthy Controls); Group 11 (RA)
Procedure: Blood Collection for PK Testing (60 minutes post injection) — Blood will be collected for subjects enrolled in Groups 10-11 for the purpose of PK analysis at 60 ± 15 minutes post injection of Tc 99m tilmanocept
  Arms: Group 10 (Healthy Controls); Group 11 (RA)
Procedure: Blood Collection for PK Testing (180 minutes post injection) — Blood will be collected for subjects enrolled in Groups 10-11 for the purpose of PK analysis at 180 ± 15 minutes post injection of Tc 99m tilmanocept
  Arms: Group 10 (Healthy Controls); Group 11 (RA)
Procedure: Blood Collection for PK Testing (18-20 hours post injection) — Blood will be collected for subjects enrolled in Groups 10-11 for the purpose of PK analysis at 18-20 hours post injection of Tc 99m tilmanocept
  Arms: Group 10 (Healthy Controls); Group 11 (RA)
Procedure: Planar Image with both Hands in Field of View — Subjects in Groups 1-9 and Groups 10 and 11 will receive planar imaging with both hands in the field of view at 60 and 180 minutes post-injection.

SUMMARY:
Prospective, open-label, multicenter, dose escalation, safety with pharmacokinetics (PK) and dosimetry study of injected Tc 99m tilmanocept in the detection of and assessment of localization to skeletal joints in subjects with and without active RA by SPECT imaging.

DETAILED DESCRIPTION:
A Manocept Platform prospective, open-label, multicenter, dose escalation, safety with PK and dosimetry study of injected Tc 99m tilmanocept in the detection of and assessment of localization to skeletal joints in subjects with and without active RA by SPECT imaging. All subjects will receive IV administration at one of 3 mass doses: 50 µg, 200 µg, or 400 µg. Within each mass dose group, subjects will receive Tc 99m tilmanocept labeled with one of 3 radiolabel doses: 1 mCi, 5 mCi, or 10 mCi.

All subjects will have a whole body planar SPECT scan. Subjects enrolled in Groups 1-9 will receive a whole body and planar hands scan followed by SPECT/CT scans on areas of interest post injection at 60 minutes ± 15 minutes and 180 minutes ± 15 minutes. Subjects enrolled in Groups 10-11 will receive a whole body planar SPECT scan performed at 4 specified time points post injection: 15 ± 5 minutes, 60 ± 15 minutes, 180 ± 15 minutes and 18-20 hours. Planar hand scans will be collected at 60 ± 15 minutes and 180 ± 15 minutes post-injection. PK blood sampling will be performed before injection (within 15 minutes), immediately following injection (within 5 minutes) and at each scanning timepoint. Dosimetry tests will be performed at each scanning timepoint. PK of urine will be assessed through counts of the bladder wall obtained from cumulative quantitative planar imaging from radiation dosimetry.

ELIGIBILITY:
Inclusion Criteria:

ALL SUBJECTS:

* The subject has provided written informed consent with HIPAA (Health Information Portability and Accountability Act) authorization before the initiation of any study-related procedures.
* Has a negative urine drug screening for illicit or unprescribed drugs suggestive of drug abuse.
* All subjects shall be ≥18 years of age at the time of consent.

CONTROL SUBJECTS:

* The subject is deemed to be clinically free of any inflammatory disease (s) and has not experienced joint pain for at least 4 weeks prior to the consent date.

ACTIVE RHEUMATOID ARTHRITIS SUBJECTS:

* The subject has moderate to severe RA as determined by the 2010 ACR/EULAR (score of ≥ 6/10).
* The subject has a DAS28 of ≥ 3.2 (includes the Erythrocyte Sedimentation Rate [ESR] test and Visual Analog Scale [VAS]) .
* If the subject is receiving methotrexate, they have been at a stable dose for > 4 weeks prior to the Baseline Visit 2 (Day 1).
* If the subject is receiving biologic therapy, they have been at a stable dose > 8 weeks prior to the Baseline Visit 2 (Day 1).
* If the subject is receiving NSAIDS or oral corticosteroids, the dose has been at a stable dose for > 4 weeks prior to the Baseline Visit 2 (Day 1). The corticosteroid dose should be ≤ 10mg/day of prednisone or an equivalent steroid dose.

Exclusion Criteria:

* The subject is pregnant or lactating.
* The subject size or weight is not compatible with imaging per the investigator.
* The subject has had or is currently receiving radiation therapy or chemotherapy for a condition other than rheumatoid arthritis.
* The subject has renal insufficiency as demonstrated by serum creatinine clearance of < 60 mL/min.
* The subject has hepatic insufficiency as demonstrated by ALT or AST greater than two times the upper limit of normal.
* The subject has a chronic or persistent infection or has any condition that would, in the opinion of the examining physician, preclude their participation.
* The subject has a known allergy to or has had an adverse reaction to dextran exposure.
* The subject has received an investigational product within 30 days prior to the Tc 99m tilmanocept administration.
* The subject has received any radiopharmaceutical within 7 days prior to the administration of Tc 99m tilmanocept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Blue, MD, Study Director — Navidea Biopharmaceuticals
Locations (1):
- Kettering Medical Center, Kettering, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 10 (Healthy Controls): Group 10 will receive the maximum tested dose of 400 mcg tilmanocept radiolabeled with 10 mCi of Tc 99m at the MTD via IV injection.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Whole body planar SPECT imaging (15 Minutes post-injection), Whole body planar SPECT imaging (60 minutes post-injection), Whole body planar SPECT imaging (180 minutes post-injection), and Whole body planar SPECT imaging (18-20 hours post-injection).
  Planar Image with both Hands in Field of View (60 minutes and 180 minutes post-injection).
  Blood Collection for PK Testing (15 Mins Before Injection), Blood Collection for PK Testing (after Injection), Blood Collection for PK Testing (15 minutes post injection), Blood Collection for PK Testing (60 minutes post injection), Blood Collection for PK Testing (180 minutes post injection), and Blood Collection for PK Testing (18-20 hours post injection).
- Group 11 (RA): Group 11 will receive the maximum tested dose of 400 mcg tilmanocept radiolabeled with 10 mCi of Tc 99m at the MTD via IV injection.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Whole body planar SPECT imaging (15 Minutes post-injection), Whole body planar SPECT imaging (60 minutes post-injection), Whole body planar SPECT imaging (180 minutes post-injection), and Whole body planar SPECT imaging (18-20 hours post-injection).
  Planar Image with both Hands in Field of View (60 minutes and 180 minutes post-injection).
  Blood Collection for PK Testing (15 Mins Before Injection), Blood Collection for PK Testing (after Injection), Blood Collection for PK Testing (15 minutes post injection), Blood Collection for PK Testing (60 minutes post injection), Blood Collection for PK Testing (180 minutes post injection), and Blood Collection for PK Testing (18-20 hours post injection).
Period: Overall Study
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 11 (RA): Group 11 will receive the maximum tested dose of 400 mcg tilmanocept radiolabeled with 10 mCi of Tc 99m the MTD via IV injection.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Whole body planar SPECT imaging (15 Minutes post-injection), Whole body planar SPECT imaging (60 minutes post-injection), Whole body planar SPECT imaging (180 minutes post-injection), and Whole body planar SPECT imaging (18-20 hours post-injection).
  Planar Image with both Hands in Field of View (60 minutes and 180 minutes post-injection).
  Blood Collection for PK Testing (15 Mins Before Injection), Blood Collection for PK Testing (after Injection), Blood Collection for PK Testing (15 minutes post injection), Blood Collection for PK Testing (60 minutes post injection), Blood Collection for PK Testing (180 minutes post injection), and Blood Collection for PK Testing (18-20 hours post injection).
- Total: Total of all reporting groups
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 39
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (8.14) | 58.7 (4.73) | 55.0 (11.16) | 46.3 (9.87) | 50.7 (12.74) | 52.0 (12.53) | 53.3 (5.69) | 56.3 (8.14) | 58.0 (3.00) | 32.0 (12.55) | 55.0 (11.16) | 54.2 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 30
  Male | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 4 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 4
  White | 2 | 2 | 2 | 3 | 3 | 1 | 2 | 2 | 1 | 3 | 5 | 26
  More than one race | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 39
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.4 (7.4) | 29.8 (3.10) | 33.5 (7.5) | 29.5 (8.47) | 39.2 (11.75) | 39.3 (8.80) | 29.2 (4.76) | 34.5 (4.62) | 33.5 (6.37) | 27.3 (7.74) | 33.5 (7.5) | 32.7 (7.72)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Drug Reaction
Description: Number of participants that experienced pharmacologic activity or ADR in each dose group.
Time Frame: From Enrollment to termination, up to 53 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6
Participants | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6

2. Secondary Outcome: Per Subject Localization Rate of Tc 99m Tilmanocept by SPECT Imaging
Description: Tc 99m Tilmanocept localization is defined as the visually (i.e., qualitatively) determined binary categorization of Tc 99m tilmanocept activity in a given DAS28 joint. The purpose of the visual assessments is to obtain dichotomized classifications of tracer uptake (herein referenced as 'localization') on planar images. Per subject localization rate is the number of subjects with at least one localized DAS28 joint per number of subjects in the analysis population.
Time Frame: For Groups 1-9, 60 ± 15 min or 180 ± 15 minute post injection planar and SPECT/CT images are used
Population: Subjects enrolled in Groups 10 and 11 received whole-body planar scans following Tc99 administration for PK and dosimetry analyses only.
Measure: Number; unit: participants
Groups:
- Group 10 (Healthy Controls): Group 10 will receive the maximum tested dose of 400 mcg tilmanocept radiolabeled with 10 mCi of Tc99m at the MTD via IV injection.
  Whole body planar SPECT imaging (15 Minutes post-injection), Whole body planar SPECT imaging (60 minutes post-injection), Whole body planar SPECT imaging (180 minutes post-injection), and Whole body planar SPECT imaging (18-20 hours post-injection)
  Planar Image with both Hands in Field of View (60 minutes and 180 minutes post-injection).
  Blood Collection for PK Testing (15 Mins Before Injection), Blood Collection for PK Testing (after Injection), Blood Collection for PK Testing (15 minutes post injection), Blood Collection for PK Testing (60 minutes post injection), Blood Collection for PK Testing (180 minutes post injection), and Blood Collection for PK Testing (18-20 hours post injection).
- Group 11 (RA): Group 11 will receive the maximum tested dose of 400 mcg tilmanocept radiolabeled with 10 mCi of Tc99m-tilmanocept at the MTD via IV injection.
  Whole body planar SPECT imaging (15 Minutes post-injection), Whole body planar SPECT imaging (60 minutes post-injection), Whole body planar SPECT imaging (180 minutes post-injection), and Whole body planar SPECT imaging (18-20 hours post-injection)
  Planar Image with both Hands in Field of View (60 minutes and 180 minutes post-injection).
  Blood Collection for PK Testing (15 Mins Before Injection), Blood Collection for PK Testing (after Injection), Blood Collection for PK Testing (15 minutes post injection), Blood Collection for PK Testing (60 minutes post injection), Blood Collection for PK Testing (180 minutes post injection), and Blood Collection for PK Testing (18-20 hours post injection).
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0
participants
  60 ± 15 min | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 |  |
  180 ± 15 min | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 |  |

3. Secondary Outcome: Tc 99m Tilmanocept Joint Localization Rate in Rheumatoid Arthritis Identified Joints
Description: Per joint (clinically RA-identified) joint localization rate of Tc 99m tilmanocept is defined as the number of localized joints per number of joints from subjects in the analysis population Groups 1-9 using SPECT imaging.
Time Frame: Whole-body planar scan at 60 ± 15 and 180 ± 15 minutes post Tc 99m tilmanocept administration with a duration of approximately 25 to 30 minutes at each timepoint.
Population: Groups 10 & 11 were not included in the population these endpoints were evaluated for.
Measure: Count of Units; unit: Joint
Units Other Than Participants: Joint
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0
Number analyzed (Joint) | 23 | 82 | 45 | 32 | 13 | 52 | 16 | 24 | 29 | 0 | 0
Joint
  Joint localization at 1 hr | 7 | 40 | 25 | 12 | 5 | 28 | 5 | 13 | 12 | 0 | 0
  Joint localization at 3 hr | 16 | 42 | 20 | 20 | 8 | 24 | 11 | 11 | 17 |  |

4. Secondary Outcome: Concordance
Description: Concordance is defined as the relationship or the presence of Tc99m localization in anatomical areas of active RA defined by clinical symptomology (defined as joint swelling (SJC) and/or tenderness (TJC) during the screening DAS28 evaluation).
Time Frame: Qualitative (i.e., visual) assessments of planar images were acquired at the 60 ± 15-minute and 180 ± 15-minute timepoints in Groups 1-9.
Population: Groups 10 & 11 were not included in the population these endpoints were evaluated for.
Measure: Count of Units; unit: Joint
Units Other Than Participants: Joint
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0
Number analyzed (Joint) | 59 | 64 | 44 | 78 | 62 | 60 | 67 | 97 | 63 | 0 | 0
Joint
  Concordance at 1 hr | 21 | 32 | 17 | 39 | 31 | 29 | 30 | 53 | 35 | 0 | 0
  Concordance at 3 hr | 38 | 32 | 27 | 39 | 31 | 31 | 37 | 44 | 28 | 0 | 0

5. Secondary Outcome: Localization Intensity
Description: Localization intensity is defined as the presence of Tc99m in each DAS28 joint and is output in tilmanocept uptake value (TUV) units, as computed using the following equation:
  〖TUV〗=ROI/BRAIN×100 where ROI = decay-corrected avg voxel intensity of the joint ROI and BRAIN =decay-corrected avg voxel intensity of the brain RR
Time Frame: Post-injection imaging at 60±15 and 180±15 min
Population: Groups 1-9 only. Groups 10 and 11 were not included.
Measure: Mean (Standard Deviation); unit: TUV
Units Other Than Participants: Joints
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0
Number analyzed (Joints) | 28 | 28 | 28 | 28 | 28 | 28 | 28 | 28 | 28 | 0 | 0
TUV
  60 ± 15 min L Shoulder | 138.9 (27.35) | 193.2 (85.82) | 188.4 (92.19) | 177.9 (64.22) | 135.0 (31.90) | 146.1 (35.54) | 177.6 (19.37) | 269.3 (238.60) | 152.7 (37.92) |  |
  60 ± 15 min R Shoulder | 156.1 (19.95) | 222.6 (113.08) | 181.2 (73.69) | 179.5 (65.66) | 145.7 (26.65) | 140.8 (12.82) | 180.1 (18.23) | 293.8 (255.64) | 184.8 (17.51) |  |
  60 ± 15 min L Elbow | 68.3 (3.38) | NA (NA) — Result from all 3 group participants not available due to joint being outside of image field of view. | 76.6 (NA) — Result from 2 of 3 group participants not available due to joint being outside of image field of view. | NA (NA) — Result from all 3 group participants not available due to joint being outside of image field of view. | NA (NA) — Result from all 3 group participants not available due to joint being outside of image field of view. | NA (NA) — Result from all 3 group participants not available due to joint being outside of image field of view. | 104.7 (22.16) | 82.3 (15.04) | 72.1 (4.87) |  |
  60 ± 15 min R Elbow | 87.4 (4.94) | 88.4 (NA) — Result from 2 of 3 group participants not available due to joint being outside of image field of view. | NA (NA) — Result from all 3 group participants not available due to joint being outside of image field of view. | 94.7 (19.29) | 76.5 (NA) — Result from 2 of 3 group participants not available due to joint being outside of image field of view. | NA (NA) — Result from all 3 group participants not available due to joint being outside of image field of view. | 110.3 (14.34) | 101.1 (16.15) | 77.3 (13.07) |  |
  60 ± 15 min L Wrist | 292.7 (96.46) | 415.9 (55.06) | 332.7 (168.46) | 416.1 (202.00) | 246.3 (109.90) | 358.4 (136.55) | 387.4 (157.13) | 472.9 (386.02) | 368.8 (146.85) |  |
  60 ± 15 min R Wrist | 387.6 (246.92) | 420.9 (59.76) | 351.3 (139.75) | 458.5 (282.25) | 271.9 (88.55) | 432.4 (268.22) | 465.5 (254.62) | 492.0 (351.80) | 337.6 (191.93) |  |
  60 ± 15 min L MCP1 | 192.2 (5.81) | 299.2 (51.36) | 203.1 (64.07) | 230.2 (97.52) | 222.9 (81.58) | 186.0 (18.29) | 241.4 (41.31) | 250.7 (95.14) | 326.9 (123.01) |  |
  60 ± 15 min L MCP2 | 175.1 (23.18) | 394.3 (152.28) | 318.7 (148.66) | 243.8 (101.78) | 177.0 (80.29) | 167.6 (43.83) | 333.5 (68.95) | 323.6 (263.03) | 248.3 (132.40) |  |
  60 ± 15 min L MCP3 | 187.1 (28.12) | 408.7 (64.48) | 259.4 (118.16) | 228.7 (123.51) | 206.7 (87.69) | 187.9 (44.78) | 286.5 (26.59) | 324.0 (258.57) | 270.5 (122.88) |  |
  60 ± 15 min L MCP4 | 181.0 (40.41) | 374.9 (103.52) | 204.7 (78.91) | 225.3 (93.15) | 214.8 (93.50) | 185.5 (50.83) | 253.1 (61.97) | 240.9 (221.84) | 211.7 (75.61) |  |
  60 ± 15 min L MCP5 | 141.9 (28.51) | 323.4 (77.01) | 159.4 (67.15) | 207.1 (87.17) | 206.5 (101.51) | 166.2 (34.36) | 236.1 (42.07) | 220.3 (152.82) | 220.9 (59.92) |  |
  60 ± 15 min R MCP1 | 238.0 (31.29) | 310.8 (41.45) | 230.0 (73.68) | 261.1 (155.97) | 254.9 (78.65) | 226.3 (57.31) | 261.6 (27.81) | 354.4 (162.04) | 349.4 (213.53) |  |
  60 ± 15 min R MCP2 | 231.7 (26.52) | 405.4 (153.35) | 285.8 (106.50) | 295.1 (227.83) | 188.6 (58.65) | 272.7 (183.37) | 286.7 (46.46) | 269.6 (167.41) | 286.1 (114.89) |  |
  60 ± 15 min R MCP 3 | 245.8 (19.43) | 353.6 (45.80) | 237.7 (135.01) | 296.9 (156.42) | 229.1 (72.37) | 234.8 (122.53) | 267.8 (44.47) | 323.9 (288.11) | 336.0 (158.66) |  |
  60 ± 15 min R MCP4 | 224.4 (20.27) | 326.4 (59.57) | 189.9 (102.96) | 231.4 (147.10) | 223.3 (78.82) | 242.7 (143.34) | 259.0 (62.48) | 265.8 (137.12) | 290.5 (133.03) |  |
  60 ± 15 min R MCP5 | 182.3 (4.68) | 316.1 (109.30) | 153.9 (85.85) | 208.0 (140.89) | 162.2 (53.15) | 192.0 (69.35) | 219.6 (86.83) | 222.1 (117.16) | 215.5 (103.57) |  |
  60 ± 15 min L PIP1 | 130.4 (5.02) | 239.3 (91.26) | 127.2 (48.94) | 196.6 (98.77) | 148.4 (53.25) | 134.8 (21.00) | 201.2 (113.75) | 166.8 (100.57) | 243.9 (14.08) |  |
  60 ± 15 min L PIP2 | 120.7 (14.68) | 158.4 (55.78) | 105.4 (49.80) | 153.3 (72.08) | 129.8 (55.88) | 126.0 (17.08) | 177.9 (18.887) | 129.9 (41.93) | 165.6 (46.37) |  |
  60 ± 15 min L PIP3 | 125.7 (7.78) | 212.3 (93.24) | 117.0 (58.62) | 170.1 (105.66) | 129.8 (65.39) | 120.2 (12.47) | 201.1 (48.49) | 204.0 (160.22) | 200.3 (85.58) |  |
  60 ± 15 min L PIP4 | 109.6 (8.41) | 172.9 (20.07) | 106.9 (43.54) | 151.8 (56.55) | 126.3 (58.40) | 117.5 (24.73) | 163.8 (53.06) | 215.6 (152.95) | 171.4 (75.27) |  |
  60 ± 15 min L PIP5 | 95.2 (14.68) | 126.3 (38.80) | 86.6 (23.94) | 138.5 (89.37) | 108.9 (66.64) | 96.4 (13.92) | 149.5 (54.15) | 215.6 (183.50) | 160.8 (36.56) |  |
  60 ± 15 min R PIP1 | 165.5 (6.81) | 285.6 (51.59) | 141.7 (71.45) | 171.3 (71.34) | 152.8 (48.86) | 148.7 (6.24) | 208.5 (39.27) | 244.8 (154.04) | 239.4 (74.89) |  |
  60 ± 15 min R PIP2 | 137.5 (12.17) | 184.6 (33.97) | 121.7 (61.52) | 194.8 (97.92) | 139.7 (56.90) | 133.3 (49.95) | 215.1 (35.17) | 198.1 (144.14) | 187.0 (77.42) |  |
  60 ± 15 min R PIP3 | 156.6 (6.02) | 189.6 (18.21) | 124.5 (74.14) | 215.0 (127.88) | 140.7 (30.08) | 168.1 (95.49) | 191.8 (43.07) | 224.3 (141.68) | 189.5 (44.79) |  |
  60 ± 15 min R PIP4 | 133.2 (19.03) | 200.5 (83.90) | 125.4 (99.16) | 161.3 (93.41) | 143.0 (53.77) | 143.6 (57.59) | 160.7 (50.81) | 221.6 (161.97) | 156.8 (47.62) |  |
  60 ± 15 min R PIP5 | 107.9 (13.12) | 174.7 (59.35) | 88.9 (54.01) | 144.3 (66.00) | 104.0 (33.68) | 104.3 (29.19) | 186.8 (36.75) | 170.9 (91.39) | 170.5 (103.26) |  |
  60 ± 15 min L Knee | 66.5 (17.79) | 107.4 (38.98) | 79.5 (18.89) | 101.4 (23.40) | 79.6 (15.84) | 78.5 (32.65) | 86.8 (14.06) | 176.7 (170.34) | 124.0 (16.81) |  |
  60 ± 15 min R Knee | 76.2 (23.25) | 118.8 (50.05) | 99.3 (36.85) | 98.3 (22.13) | 78.7 (14.07) | 67.1 (8.62) | 91.1 (14.44) | 165.4 (174.57) | 133.7 (22.82) |  |
  180 ± 15 min L Shoulder | 165.4 (54.95) | 210.1 (89.77) | 232.2 (116.41) | 211.0 (81.71) | 160.8 (55.63) | 163.0 (37.4) | 218.0 (67.76) | 301.4 (254.58) | 181.4 (66.68) |  |
  180 ± 15 min R Shoulder | 189.1 (51.36) | 240.5 (118.56) | 230.0 (81.69) | 209.3 (86.04) | 177.6 (54.82) | 148.9 (12.60) | 221.6 (59.4) | 321.0 (237.86) | 206.1 (41.31) |  |
  180 ± 15 min L Elbow | 71.8 (13.49) | NA (NA) — Result from all 3 group participants not available due to joint being outside of image field of view. | 76.2 (NA) — Result from 2 of 3 group participants not available due to joint being outside of image field of view. | 102.4 (49.11) | 57.7 (NA) — Result from 2 of 3 group participants not available due to joint being outside of image field of view. | NA (NA) — Result from all 3 group participants not available due to joint being outside of image field of view. | 94.6 (13.84) | 101.2 (25.92) | 91.0 (2.59) |  |
  180 ± 15 min R elbow | 85.5 (7.77) | 97.3 (NA) — Result from 2 of 3 group participants not available due to joint being outside of image field of view. | 85.9 (NA) — Result from 2 of 3 group participants not available due to joint being outside of image field of view. | 109.3 (44.46) | 71.2 (NA) — Result from 2 of 3 group participants not available due to joint being outside of image field of view. | NA (NA) — Result from all 3 group participants not available due to joint being outside of image field of view. | 102.1 (28.42) | 94.3 (4.39) | 90.9 (5.49) |  |
  180 ± 15 min L Wrist | 401.8 (201.69) | 488.6 (40.47) | 434.0 (183.81) | 514.7 (275.68) | 299.7 (126.01) | 404.1 (126.88) | 457.9 (157.64) | 566.6 (374.43) | 484.7 (164.36) |  |
  180 ± 15 min R Wrist | 387.6 (246.92) | 479.7 (73.26) | 482.2 (169.64) | 582.1 (411.89) | 404.5 (177.65) | 465.1 (269.97) | 565.6 (283.40) | 534.7 (314.36) | 456.8 (194.99) |  |
  180 ± 15 min L MCP1 | 527.8 (355.31) | 309.9 (57.82) | 293.9 (93.47) | 321.2 (169.11) | 300.3 (136.28) | 216.6 (17.24) | 259.7 (56.52) | 297.4 (107.98) | 327.7 (58.96) |  |
  180 ± 15 min L MCP2 | 259.7 (67.37) | 378.4 (212.17) | 404.1 (168.75) | 316.1 (114.50) | 252.7 (139.89) | 225.7 (30.86) | 300.6 (157.04) | 364.3 (184.71) | 237.1 (131.01) |  |
  180 ± 15 min L MCP3 | 252.3 (60.46) | 456.5 (90.38) | 327.1 (97.70) | 317.3 (184.41) | 302.4 (146.85) | 220.4 (63.17) | 393.1 (57.80) | 364.2 (210.61) | 300.5 (84.15) |  |
  180 ± 15 min L MCP4 | 219.8 (44.10) | 414.3 (76.72) | 273.5 (71.29) | 278.8 (139.18) | 261.5 (128.77) | 195.4 (39.10) | 361.9 (60.33) | 315.2 (195.40) | 305.5 (97.92) |  |
  180 ± 15 min L MCP5 | 179.8 (59.65) | 413.1 (81.96) | 203.2 (61.46) | 264.4 (165.09) | 251.9 (128.70) | 184.4 (44.55) | 276.4 (62.35) | 298.0 (104.10) | 228.8 (43.52) |  |
  180 ± 15 min R MCP1 | 298.9 (68.07) | 344.3 (25.68) | 284.4 (68.47) | 351.1 (222.79) | 288.4 (127.85) | 258.6 (71.85) | 346.9 (33.49) | 356.0 (64.44) | 416.8 (194.14) |  |
  180 ± 15 min R MCP2 | 289.9 (37.14) | 495.1 (256.02) | 341.6 (126.66) | 405.0 (343.20) | 271.4 (146.89) | 300.3 (147.97) | 294.3 (40.20) | 397.0 (170.33) | 340.5 (169.41) |  |
  180 ± 15 min R MCP3 | 320.9 (76.70) | 428.1 (5.42) | 286.9 (118.06) | 404.0 (242.78) | 300.1 (171.48) | 298.2 (138.42) | 330.5 (97.94) | 385.2 (256.76) | 367.9 (121.03) |  |
  180 ± 15 min R MCP4 | 263.6 (24.44) | 380.8 (38.83) | 271.1 (101.92) | 320.0 (202.62) | 284.2 (137.20) | 271.2 (73.89) | 255.3 (56.27) | 361.8 (223.67) | 363.7 (104.49) |  |
  180 ± 15 min R MCP5 | 214.5 (37.25) | 373.2 (122.41) | 218.4 (67.7) | 276.1 (168.15) | 262.1 (140.52) | 187.3 (34.76) | 270.6 (58.95) | 332.5 (162.83) | 369.2 (77.77) |  |
  180 ± 15 min L PIP1 | 179.4 (41.32) | 270.7 (98.35) | 177.0 (76.74) | 220.4 (125.71) | 224.0 (146.46) | 156.1 (8.23) | 206.3 (25.63) | 275.1 (74.03) | 254.3 (95.16) |  |
  180 ± 15 min L PIP2 | 144.4 (12.55) | 165.9 (44.85) | 151.2 (38.91) | 209.8 (116.11) | 189.5 (106.68) | 142.4 (18.60) | 227.5 (50.02) | 285.4 (229.72) | 204.8 (63.14) |  |
  180 ± 15 min L PIP3 | 152.4 (45.18) | 257.6 (126.40) | 157.8 (72.64) | 215.3 (120.83) | 160.7 (81.29) | 155.2 (54.09) | 224.2 (5.85) | 285.6 (241.39) | 204.4 (84.03) |  |
  180 ± 15 min L PIP4 | 133.6 (22.67) | 185.2 (10.12) | 150.9 (48.91) | 195.7 (120.38) | 167.2 (96.27) | 157.8 (28.39) | 249.7 (77.85) | 246.4 (191.83) | 198.6 (85.67) |  |
  180 ± 15 min L PIP5 | 104.1 (17.04) | 151.0 (25.51) | 124.2 (27.15) | 191.1 (149.39) | 143.7 (98.53) | 109.1 (16.35) | 219.4 (95.36) | 183.6 (85.21) | 168.3 (58.47) |  |
  180 ± 15 min R PIP1 | 218.6 (53.24) | 309.0 (60.52) | 202.1 (67.80) | 221.3 (133.90) | 222.0 (117.48) | 194.1 (32.36) | 303.2 (62.42) | 261.8 (138.92) | 262.7 (83.66) |  |
  180 ± 15 min R PIP2 | 193.0 (43.56) | 204.7 (18.16) | 174.8 (67.84) | 256.4 (140.51) | 187.3 (75.12) | 164.9 (57.27) | 211.9 (56.41) | 200.5 (47.74) | 225.4 (9.65) |  |
  180 ± 15 min R PIP3 | 182.4 (14.8) | 224.8 (21.69) | 164.0 (64.36) | 239.6 (135.40) | 184.9 (76.62) | 198.0 (85.74) | 255.0 (65.78) | 263.1 (120.11) | 229.3 (44.24) |  |
  180 ± 15 min R PIP4 | 164.6 (30.74) | 376.6 (103.08) | 175.3 (78.67) | 213.4 (147.22) | 170.3 (97.90) | 182.8 (47.32) | 243.5 (36.60) | 292.8 (174.85) | 196.2 (108.71) |  |
  180 ± 15 min R PIP5 | 125.7 (8.97) | 200.3 (73.56) | 119.7 (30.65) | 181.4 (90.31) | 148.5 (64.16) | 117.3 (44.55) | 147.5 (47.18) | 233.4 (102.14) | 197.7 (50.77) |  |
  180 ± 15 min L Knee | 80.5 (26.70) | 113.8 (39.80) | 104.5 (27.67) | 126.1 (43.18) | 98.6 (25.98) | 87.5 (37.21) | 101.2 (32.64) | 193.7 (177.10) | 146.8 (22.71) |  |
  180 ± 15 min R Knee | 92.5 (39.11) | 126.5 (47.90) | 124.0 (40.28) | 122.1 (40.79) | 105.3 (23.75) | 76.5 (11.68) | 107.5 (37.05) | 191.4 (180.37) | 151.8 (25.49) |  |

6. Secondary Outcome: Per Subject Localization Rate of Tc 99m Tilmanocept in Areas Other Than RA
Description: Per subject localization rate of Tc 99m tilmanocept in areas other than RA is defined as the number of subjects with at least one localized DAS28 joint per number of subjects in the analysis population.
Time Frame: Imaging taken 60 ± 15 min and 180 ± 15 min post-injection
Population: Only Groups 1-9. Groups 10 & 11 were not included in the population these endpoints were evaluated for.
Measure: Number; unit: participants
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0
participants
  Number of subjects localized at 60 ± 15 min | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 |  |
  Number of subjects localized at 180 ± 15 min | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 |  |

7. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: Maximum observed concentration (Cmax) will be calculated, whenever possible, using Tc 99m tilmanocept total radioactivity in whole blood and urine.
Time Frame: 15 minutes prior to administration. Immediately after administration. 15 ± 5 minutes post administration • 60 ± 15 minutes post administration • 180 ± 15 minutes post administration • 18 to 20 hours post administration
Population: Only in Groups 10 and 11
Measure: Mean (90% Confidence Interval); unit: nCi/mL
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
nCi/mL |  |  |  |  |  |  |  |  |  | 1244.2 [809.55 to 1649.33] | 2043.8 [1078.28 to 2878.94]

8. Secondary Outcome: Time to Cmax (Tmax)
Description: Time to Cmax (tmax) will be calculated, whenever possible, using Tc 99m tilmanocept total radioactivity in whole blood and urine.
Time Frame: Radioactivity was quantitated at each time point -15 mins prior to administration• Immediately after administration •15 ± 5 minutes post administration • 60 ± 15 minutes post administration • 180 ± 15 minutes post administration • 18 to 20 hours post admi
Population: Groups 10 and 11
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
minutes |  |  |  |  |  |  |  |  |  | 27.3 (7.36) | 255 (6.58)

9. Secondary Outcome: Area Under the Concentration-time Curve (AUC) From Hour 0 to the Last Measureable Concentration (AUC0-t)
Description: Area under the concentration-time curve (AUC) from Hour 0 to the last measureable concentration (18 to 20 hours) (AUC0-t) will be calculated, whenever possible, using Tc 99m tilmanocept total radioactivity in whole blood and urine.
Time Frame: Hour 0 to hour 18-20, with time points immediately post injection, 0.25 hr, 1 hr, 3 hr and 18-20 hr after injection
Population: Groups 10 and 11
Measure: Mean (90% Confidence Interval); unit: min*nCi/mL
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
min*nCi/mL
  Whole blood AUC |  |  |  |  |  |  |  |  |  | 235258.0 [193698.75 to 275134.27] | 268110.7 [217187.41 to 316806.03]
  Urine AUC |  |  |  |  |  |  |  |  |  | 1468788.9 [1088888.09 to 1830437.75] | 1384642.0 [1123310.11 to 1634810.07]

10. Secondary Outcome: AUC Extrapolated to Infinity
Description: AUC extrapolated to infinity will be calculated, whenever possible, using Tc 99m tilmanocept total radioactivity in whole blood and urine.
Time Frame: 15 mins prior to administration • Immediately after administration • 15 ± 5 minutes post administration • 60 ± 15 minutes post administration • 180 ± 15 minutes post administration • 18 to 20 hours post administration
Population: Groups 10 and 11 only.
Measure: Mean (90% Confidence Interval); unit: min*nCi/mL
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
min*nCi/mL |  |  |  |  |  |  |  |  |  | 370580.1 [290005.04 to 447777.17] | 396026.4 [315475.79 to 472251.44]

11. Secondary Outcome: Apparent Terminal Elimination Rate Constant (Z)
Description: Apparent terminal elimination rate constant (Z) will be calculated, whenever possible, using Tc 99m tilmanocept total radioactivity in whole blood and urine.
Time Frame: as for outcome 10
Population: Groups 10 and 11 only.
Measure: Mean (90% Confidence Interval); unit: 1/minute
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
1/minute |  |  |  |  |  |  |  |  |  | 0.00094 [0.00080 to 0.00107] | 0.00100 [0.00083 to 0.00116]

12. Secondary Outcome: Apparent Terminal Elimination Half-life (t1/2)
Description: Apparent terminal elimination half-life (t1/2) will be calculated, whenever possible, using Tc 99m tilmanocept total radioactivity in whole blood and urine.
Time Frame: as for outcome 10
Population: Groups 10 and 11.
Measure: Mean (90% Confidence Interval); unit: minutes
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
minutes |  |  |  |  |  |  |  |  |  | 759.0 [648.36 to 865.85] | 719.1 [598.97 to 835.46]

13. Secondary Outcome: Radiation Dosimetry of Tc 99m Tilmanocept
Description: Mean total radiation dose per organ (mSv/MBq) in HC females, HC males, females with active RA, and males with active RA.
  Results were obtained at the subject level from Hybrid Dosimetry™ Version 2.8.3 and OLINDA/EXM® Version 2.1RC93 in accordance with NAV3-21 Protocol Amendment 6. The Hybrid Dosimetry™ function provides an efficient way to generate kinetic data for selected organs via regions of interest (ROI) drawing. From this data, residence times are calculated and transferred to OLINDA/EXM®, which generates absorbed dose tables using the MIRD methodology.
Time Frame: Planar images were taken 15 ± 5 minutes, 60 ± 5 minutes, 180 ± 5 minutes, 18 to 20 hours after Tc 99m tilmanocept administration and processed in accordance with the NAV3-21 protocol endpoints using established dosimetry software.
Population: Groups 10 and 11 will receive the maximum tested dose of 400 mcg tilmanocept radiolabeled with 10 mCi of Tc 99m at the MTD via IV injection.
Measure: Mean (Standard Deviation); unit: mSv/MBq
Groups:
- Group 10 (HC Females): Group 10 will receive the maximum tested dose of 400 mcg tilmanocept radiolabeled with 10 mCi of Tc 99m at the MTD via IV injection.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Whole body planar SPECT imaging (15 Minutes post-injection), Whole body planar SPECT imaging (60 minutes post-injection), Whole body planar SPECT imaging (180 minutes post-injection), and Whole body planar SPECT imaging (18-20 hours post-injection).
  Planar Image with both Hands in Field of View (60 minutes and 180 minutes post-injection).
  Blood Collection for PK Testing (15 Mins Before Injection), Blood Collection for PK Testing (after Injection), Blood Collection for PK Testing (15 minutes post injection), Blood Collection for PK Testing (60 minutes post injection), Blood Collection for PK Testing (180 minutes post injection), and Blood Collection for PK Testing (18-20 hours post injection).
- Group 10 (HC Males); Group 11 (RA Females); Group 11 (RA Males): Group 11 will receive the maximum tested dose of 400 mcg tilmanocept radiolabeled with 10 mCi of Tc 99m at the MTD via IV injection.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Whole body planar SPECT imaging (15 Minutes post-injection), Whole body planar SPECT imaging (60 minutes post-injection), Whole body planar SPECT imaging (180 minutes post-injection), and Whole body planar SPECT imaging (18-20 hours post-injection).
  Planar Image with both Hands in Field of View (60 minutes and 180 minutes post-injection).
  Blood Collection for PK Testing (15 Mins Before Injection), Blood Collection for PK Testing (after Injection), Blood Collection for PK Testing (15 minutes post injection), Blood Collection for PK Testing (60 minutes post injection), Blood Collection for PK Testing (180 minutes post injection), and Blood Collection for PK Testing (18-20 hours post injection).
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (HC Females) | Group 10 (HC Males) | Group 11 (RA Females) | Group 11 (RA Males)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3
mSv/MBq |  |  |  |  |  |  |  |  |  | 4.69 (4.54) | 2.69 (1.13) | 5.06 (4.93) | 3.02 (2.97)

ADVERSE EVENTS:
Time Frame: 53 days
Arm/Group | Group 1 (RA) | Group 2 (RA) | Group 3 (RA) | Group 4 (RA) | Group 5 (RA) | Group 6 (RA) | Group 7 (RA) | Group 8 (RA) | Group 9 (RA) | Group 10 (Healthy Controls) | Group 11 (RA)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 0/3 | 0/3 | 0/3 | 0/3 | 1/3 | 0/3 | 1/3 | 0/3 | 2/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (RA) (N=3) | Group 2 (RA) (N=3) | Group 3 (RA) (N=3) | Group 4 (RA) (N=3) | Group 5 (RA) (N=3) | Group 6 (RA) (N=3) | Group 7 (RA) (N=3) | Group 8 (RA) (N=3) | Group 9 (RA) (N=3) | Group 10 (Healthy Controls) (N=6) | Group 11 (RA) (N=6)
Hypoglycemia (Endocrine disorders) | 0 | 0 | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Fatigue (General disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and make modifications to the publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT02865434/Prot_SAP_000.pdf